CLINICAL TRIAL: NCT04834882
Title: Burnout, Stress and Coping Strategies: Impact of the Covid-19 Epidemic on the Medical and Paramedical Staff in Reims University Hospital and EPSM Marne
Brief Title: Burnout, Stress and Coping Strategies: Impact of the Covid-19 Epidemic
Acronym: Au20-15
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO20152*
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Burnout, Professional
MeSH Terms: conditions — COVID-19; Burnout, Professional | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Medical and paramedical staff in Reims University Hospital and EPSM Marne working in COVID-19 units and non COVID-19 units
  Interventions: Other: Data collection (

INTERVENTIONS:
Other: Data collection ( — online survey

SUMMARY:
Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) is a novel coronavirus detected in Wuhan, China on December 2019. This virus is responsible for the infectious respiratory disease called Covid-19.

The psychological effects of this epidemic are found among the general population, but also healthcare workers. Some studies have shown that psychological disorders such as stress, anxiety, depressive symptoms, insomnia, denial, anger and fear, post-traumatic stress disorder are emerging among healthcare workers. However, there is currently insufficient data to evaluate the burnout during the COVID-19 pandemic.

The purpose of this study is to understand the impact of the covid-19 epidemic on stress and burnout on healthcare workers and their coping strategies.

DETAILED DESCRIPTION:
Burnout syndrome, a state of professional exhaustion, is prevalent among the medical and paramedical staff. The covid-19 pandemic may generate more stress and increase the risk for burnout.

The aim of this study is to evaluate burnout (prevalence and intensity) and stress of among healthcare workers in COVID-19 units and non COVID-19 units. We also explore the supportive coping strategies need to reduce their stress and burnout.

ELIGIBILITY:
Inclusion Criteria:

* Medical (physicians, interns) and paramedical (nursing managers, nurses, care assistants) staff in Reims University Hospital and EPSM Marne
* Person who have attained majority
* Person consenting to participate to the study

Exclusion Criteria:

* Healthcare workers outside of Reims University Hospital and EPSM Marne
* Person who is not a healthcare professional

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All healthcare workers participating will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Assessment of burnout (prevalence and intensity) | Day 0
  Self-Administered Questionnaires : Maslash Burnout Inventory-Human Services Survey
Assessment of stress | Day 0
  Self-Administered Questionnaires : Perceived Stress Scale

SECONDARY OUTCOMES:
Assessment of supportive coping strategies | Day 0
  Self-Administered Questionnaires : Ways of Coping Checklist (WCC-R)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided